CLINICAL TRIAL: NCT02237937
Title: Optimizing Antidepressant Treatment by Genotype-dependent Adjustment of Medication According to the ABCB1 Gene
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: HolsboerMaschmeyer NeuroChemie GmbH (Industry)
Collaborators: Max-Planck-Institute of Psychiatry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double
Other Study IDs: 2011-003190-29
Record Dates: First submitted 2013-08-26; First posted 2014-09-12 (Estimated); Last update posted 2014-09-12 (Estimated); Status verified 2014-09

CONDITIONS: Major Depression
Keywords: Depression, Affective Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Depression; Mood Disorders | interventions — Paroxetine; Sertraline; Citalopram; Venlafaxine Hydrochloride; Amitriptyline; Escitalopram; amitriptyline N-oxide; Nortriptyline; Trimipramine

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Normal dosage (Experimental): Selected antidepressants that are substrates of the P-glycoprotein:
  Dosage:
  * paroxetine < 40 mg/d
  * sertraline < 100 mg/d
  * citalopram < 40 mg/d
  * escitalopram < 20 mg/d
  * venlafaxine < 225 mg/d
  * amitriptyline < 150 mg/d
  * amitriptylinoxide < 150 mg/d
  * nortriptyline < 150 mg/d
  * trimipramine < 150 mg/d
  Interventions: Drug: Paroxetine; Drug: Sertraline; Drug: Citalopram; Drug: Venlafaxine; Drug: Amitriptyline; Drug: Escitalopram; Drug: Amitriptylinoxide; Drug: Nortriptyline; Drug: Trimipramine
- High dosage (Experimental): Selected antidepressants that are substrates of the P-glycoprotein:
  Dosage:
  * paroxetine < 80 mg/d
  * sertraline < 200 mg/d
  * citalopram < 80 mg/d
  * escitalopram < 40 mg/d
  * venlafaxine < 450 mg/d
  * amitriptyline < 300 mg/d
  * amitriptylinoxide < 300 mg/d
  * nortriptyline < 300 mg/d
  * trimipramine < 300 mg/d
  Interventions: Drug: Paroxetine; Drug: Sertraline; Drug: Citalopram; Drug: Venlafaxine; Drug: Amitriptyline; Drug: Escitalopram; Drug: Amitriptylinoxide; Drug: Nortriptyline; Drug: Trimipramine

INTERVENTIONS:
Drug: Paroxetine
Drug: Sertraline
Drug: Citalopram
Drug: Venlafaxine
Drug: Amitriptyline
Drug: Escitalopram
Drug: Amitriptylinoxide
Drug: Nortriptyline
Drug: Trimipramine

SUMMARY:
The study evaluates the ABCB1-genotype dependent efficacy of a quick dose-escalation strategy within 28 days of treatment with approved antidepressants that are known substrates of the P-glycoprotein, an efflux pump of the blood-brain barrier expressed by the ABCB1 gene.

Moreover, the study evaluates ABCB1-genotype dependent side-effects of approved antidepressants that are known substrates of the P-glycoprotein, an efflux pump of the blood-brain barrier expressed by the ABCB1 gene.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients
* Age between 18 and 80 years
* Inpatients with a DSM-IV diagnosis of Major Depression
* single episode or recurrent
* moderate to severe intensity
* without psychotic features
* Inpatients with a DSM-IV diagnosis of bipolar disorder I or II
* current episode with depressive symptoms
* moderate to severe intensity
* without psychotic features
* HAM-D score at the time of inclusion in the study ≥ 14
* Patient has already been adjusted to one of the following antidepressants in a dose which is still under the defined normal-dose:
* paroxetine < 40 mg/d
* sertraline < 100 mg/d
* citalopram < 40 mg/d
* escitalopram < 20 mg/d
* venlafaxine < 225 mg/d
* amitriptyline < 150 mg/d
* amitriptylinoxide < 150 mg/d
* nortriptyline < 150 mg/d
* trimipramine < 150 mg/d

Exclusion Criteria:

* Acute suicidality (HAM-D Item 3 score > 2)
* Acute alcohol-, hypnotics-, analgesics- or psychopharmacological intoxication or delirium
* Current alcohol dependence, or dependencies from other psychotropic substances
* Severe medical or neurological diseases: patients with severe hepatic (severe impairment of liver function, cirrhosis of the liver), renal (kidney malfunctions), cardiovascular (recent myocardial infarction, instable heart disease), neurological diseases (e.g. multiple sclerosis, Parkinson, dementia)
* Patients incapable of giving informed consent
* Pregnant or breast-feeding women
* Women of reproductive age without effective contraception
* Simultaneous participation in other clinical trials or participation in an other clinical trial within 6 weeks before the start of the study
* Hypersensitivity to the study medication or to one of the ingredients of the medication
* Simultaneous treatment with another antidepressant besides study medication (exception: trazodone up to 75 mg/d, mirtazapine up to 15 mg/d, trimipramine up to 50 mg/d)
* Simultaneous treatment with mood stabilizers or neuroleptic drugs (exception: quetiapine up to 50 mg/d, olanzapine up to 5 mg/d)
* Exclusion criteria of the study medication

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2011-09; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
25% improvement in the HAM-D | after 28 days of treatment
  Partial response indicated by at least 25% improvement in the Hamilton Rating Scale for Depression (HAM-D)

SECONDARY OUTCOMES:
side effects | after 28 days of treatment
  UKU side effect scale, AMDP side effect scale

CONTACTS AND LOCATIONS:
Overall Officials: Florian Holsboer, MD, PHD, Principal Investigator — Max-Planck-Institute of Psychiatry
Locations (1):
- Max Planck Institute of Psychiatry, Munich, Bavaria, Germany